CLINICAL TRIAL: NCT03768206
Title: Promoting Physical Activity Via Physical Therapist Following Knee Replacement- The PATH Study
Brief Title: The PATH Study to Promote Physical Activity After Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081254
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Knee Arthroplasty
Keywords: knee arthroplasty; behavioral intervention; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH (Experimental): PATH participants will receive Standard Outpatient Physical Therapy. In addition, physical therapist discuss physical activity & assist with goal setting during therapy sessions.
  Interventions: Behavioral: Standard Physical Therapy; Behavioral: Physical therapist discuss aerobic physical activity
- PATH-12 (Active Comparator): PATH-12 participants will receive Standard Outpatient Physical Therapy. In addition, PATH-12 participants will receive a Physical activity session (1-hour) focusing on physical activity and goal setting at 12 weeks after surgery.
  Interventions: Behavioral: Standard Physical Therapy; Behavioral: Physical activity session

INTERVENTIONS:
Behavioral: Standard Physical Therapy — Participants will receive standard outpatient physical therapy that is typical following knee replacement
Behavioral: Physical therapist discuss aerobic physical activity — Physical therapists will provide recommendations to increase aerobic physical activity and set goals during standard physical therapy sessions after knee replacement.
  Arms: PATH
Behavioral: Physical activity session — Participants will receive a one hour coaching session on aerobic physical activity and goal setting after knee replacement.
  Arms: PATH-12

SUMMARY:
The purpose of this study is to examine the feasibility and preliminary efficacy of a physical therapist led physical activity intervention for knee replacement patients within an outpatient physical therapy facility.

DETAILED DESCRIPTION:
Physical activity does not typically increase after knee replacement; thus, the purpose of this study is to examine if physical activity levels will be higher among knee replacement patients who receive a physical therapist led physical activity intervention during standard physical therapy sessions. Physical activity levels will be assessed at the start of outpatient therapy and at 12 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be 40-79 years of age
* Have had a knee replacement in the last 2 months
* Be willing to wear and accelerometer for 7 days during assessments
* Be English speaking

Exclusion Criteria:

* Have any contraindications to activity
* Have a mobility limiting comorbidity
* Have a scheduled surgery within the next 6 months

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, phD, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Palmetto Health- USC Orthopedic Center, Columbia, South Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No
Given the preliminary nature of the study and small sample size, we do not plan to share data with others, unless requested to do so.

REFERENCES:
- [Derived] Pellegrini CA, Brown D, DeVivo KE, Lee J, Wilcox S. Promoting physical activity via physical therapist following knee replacement: A pilot randomized controlled trial. PM R. 2023 Aug;15(8):965-975. doi: 10.1002/pmrj.12895. Epub 2022 Dec 15. PMID 36106651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PATH | PATH-12
Started | 24 | 21
Completed | 22 | 19
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PATH | PATH-12 | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (5.4) | 63.3 (8.1) | 65.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 18 | 13 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45
Moderate-vigorous intensity physical activity [Mean (Standard Deviation); unit: minutes/week] — Population: Participants were only included if they had 4 valid days of at least 10 hours of wear time
  minutes/week
    number analyzed (Participants) | 22 | 17 | 39
    (all) | 37.8 (56.8) | 23.5 (22.3) | 31.5 (45.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled
Description: Feasibility will be determined based on the number of participants enrolled vs. the number approached
Time Frame: Baseline
Population: The overall number of participants analyzed reflects the total number of participants that were approached and screened for participation
Measure: Count of Participants; unit: Participants
Groups:
- Total Participants Approached: The total number of participants that were screened for participation in the study
Arm/Group | Total Participants Approached
Number analyzed (Participants) | 136
Participants | 45

2. Primary Outcome: Percentage of Participants Who Complete the 12 Week Assessment
Description: Acceptability will be determined by the percentage of participants completing the 12 week assessment.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PATH | PATH-12
Number analyzed (Participants) | 24 | 21
Participants | 22 | 19

3. Secondary Outcome: Moderate-Vigorous Intensity Physical Activity
Description: Total number of minutes of objectively-measured moderate-vigorous intensity (>2020 counts/min) physical activity/week assessed using Actigraph link activity monitors worn around the waist for 7 days.
Time Frame: 12 weeks
Population: Only participants with 4 valid days of activity monitor wear (at least 10 hours of wear time) were included in analyses
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | PATH | PATH-12
Number analyzed (Participants) | 20 | 18
minutes/week | 48.5 (55.4) | 57.4 (62.9)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | PATH | PATH-12
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03768206/Prot_SAP_000.pdf